CLINICAL TRIAL: NCT05840796
Title: To Explore the Anti-oxidative Effects and Inflammation Effects of Soy Protein to Renal Function of End Stage Diabetes Nephropathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTMHH-103006
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- soy protein drink (Experimental): The calories oral nutrition supplements were 100 kcal, which included 8.4g of protein and phosphorous was excluded in two oral nutrition supplements formula.
  Each participant had two packs of nutrition supplement per day.
  Interventions: Dietary Supplement: soy protein drink
- casein protein drink (Other): The calories oral nutrition supplements were 100 kcal, which included 8.4g of protein and phosphorous was excluded in two oral nutrition supplements formula.
  Each participant had two packs of nutrition supplement per day.
  Interventions: Dietary Supplement: casein protein drink

INTERVENTIONS:
Dietary Supplement: soy protein drink — The calories oral nutrition supplements were 100 kcal, which included 8.4g of protein and phosphorous was excluded in two oral nutrition supplements formula.
  Each participant had two packs of nutrition supplement per day for 4months. The 24-h dietary record, blood pressure, plasma glucose, lipid profile, renal function (estimated glomerular filtration rate, eGFR), inflammatory factor levels were analyzed at the baseline and at the 4th month of the study.
  The participants were followed up until the 7th month of the study.
  Arms: soy protein drink
Dietary Supplement: casein protein drink — The calories oral nutrition supplements were 100 kcal, which included 8.4g of protein and phosphorous was excluded in two oral nutrition supplements formula.
  Each participant had two packs of nutrition supplement per day for 4 months. The 24-h dietary record, blood pressure, plasma glucose, lipid profile, renal function (estimated glomerular filtration rate, eGFR), inflammatory factor levels were analyzed at the baseline and at the 4th month of the study.
  The participants were followed up until the 7th month of the study.
  Arms: casein protein drink

SUMMARY:
This study investigated the beneficial effects of soybean on the renal function, oxidative stress, and inflammatory responses in patients with end-stage diabetic nephropathy (DN).

DETAILED DESCRIPTION:
DN outpatients were recruited from Tung's Taichung MetroHarbor Hospital (Taichung City, Taiwan). They were randomly separated into two groups; one group was given soy protein drink and the other group was given casein drink for 4 months. The blood pressure, plasma glucose, lipid profile, renal function (estimated glomerular filtration rate, eGFR), inflammatory factor levels were analyzed at the baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged from 40 to 75 years and were at DN stage 4 or 5 were enrolled in this study.

Exclusion Criteria:

* The exclusion criteria were having hemodialysis, lactose intolerance, gastrointestinal (GI) tract dysfunction, liver disease, acute metabolic acidosis or ketoacidosis, in acute infection, severe dehydration, alcohol abuse, addictive drug abuse, cancer in recent 5 years, being involved in another trial in past 1 month, had operation in the past 4 months, or had compliance lower than 90% in the first month of study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2015-02-28 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
24-hours dietary recall | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  Estimated by registered dietitian to understand calories, protein and nutrients intake..
estimated glomerular filtration rate (eGFR) | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  renal function
creatinine | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  renal function
plasma malondialdehyde (MDA) | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  Antioxidative statement-lipid peroxidation
high-sensitivity C-reactive protein (hs-CRP) | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  inflammatory indicators
soluble intercellular adhesion molecule (sICAM)-1 | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  inflammatory indicators
soluble vascular cell adhesion molecule (sVICAM)-1 | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  inflammatory indicators
interleukin (IL)-6 | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  inflammatory indicators

SECONDARY OUTCOMES:
Blood pressure | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  systolic blood pressure (SBP), diastolic blood pressure (DBP)
body weight | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  body weight
blood glucose | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  fasting plasma glucose (FPG)
lipid profile | Change from Baseline and 4th and 7th week, the intervention will last for 4 months and follow up for 3 months
  triglycerides (TG), total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C)